CLINICAL TRIAL: NCT02743520
Title: Early Identification of Patients With Coexisting Atrial Fibrillation and Obstructive Sleep Apnea
Brief Title: Arrhythmia Detection In Obstructive Sleep Apnea (ADIOS)
Acronym: ADIOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Alberto Rafael Ramos, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20150860
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation; Arrhythmia; Stroke, Cardiovascular
Keywords: sleep apnea; arrhythmia detection
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Myocardial Infarction; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cardiac event monitor (Experimental): Participants will under go evaluation with a two week cardiac event monitor.
  Interventions: Device: The Lifestar Act III

INTERVENTIONS:
Device: The Lifestar Act III — The Lifestar Act III is a chest-worn continuous Electrocardiogram (ECG) monitor and arrhythmia detector. The device is equipped with four electrodes on a harness with a Bluetooth transceiver and a buzzer. The ECG signals will be transmitted via Bluetooth to an application arranged to process and transmit the ECG recordings.

SUMMARY:
The purpose of this research study is to learn about arrhythmia detection in obstructive sleep apnea (OSA). For several years patients with OSA have an increased likelihood of having irregular heartbeats. This study will determine how often patients with OSA have irregular heartbeats. This study will also define which OSA patients are most likely to have irregular heartbeats.

The participant is being asked to be in the study because the participant has been diagnosed with obstructive sleep apnea (OSA).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of OSA within the last 12 months
2. No previous diagnosis of atrial fibrillation
3. Able and willing to follow-up as an outpatient
4. Age 40-85 years

Exclusion Criteria:

1. Life expectancy < 2 years
2. Dementia or other neurologic condition which would make outpatient follow-up difficult
3. CHADS score <2
4. Alcohol or drug abuse which would interfere with outpatient follow-up
5. Severe Congestive heart failure (NYHA class 3 or 4) or use of left ventricular assist device.
6. Current dialysis treatment or planned treatment within 12 months
7. Known bleeding disorder or prothrombin time >15 seconds
8. Mechanical heart valve requiring anticoagulation
9. Moderate to severe mitral stenosis or regurgitation
10. Prior clinical diagnosis of ischemic stroke (radiologic infarcts are not excluded)
11. Chronic obstructive pulmonary disease with oxygen dependence
12. Pregnant patients or patients that plan to become pregnant within the course of the study*.
13. Patients with anticipated need for a pacemaker during the course of the study *If any patients become pregnant during the course of the study, pregnancy outcomes will not be followed

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto R Ramos, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardiac Event Monitor
Started | 86
Completed | 85
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cardiac Event Monitor
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 63
  More than one race | 2
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Definite Atrial Fibrillation (Defined as an Irregularly Irregular Rhythm With Absence of p Waves)
Description: New cases of atrial fibrillation as evaluated by the LifestarAct III.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Event Monitor
Number analyzed (Participants) | 85
Participants | 2

2. Secondary Outcome: Number of Participants With Frequent Ventricular Premature Contractions
Description: More than 100 contraction during a 24 hour period as evaluated by the LifestarAct III.
Time Frame: week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Event Monitor
Number analyzed (Participants) | 85
Participants | 22

3. Secondary Outcome: Longest Duration of Atrial Fibrillation
Description: Longest duration of Atrial Fibrillation in minutes compare to the rests of Atrial Fibrillation in a 24 hours, as evaluated by the LifestarAct III.
Time Frame: Week 2
Population: Due to software error, data could not be extracted for analysis for this outcome for all participants
Arm/Group | Cardiac Event Monitor
Number analyzed (Participants) | 0

4. Secondary Outcome: Atrial Fibrillation Episodes Lasting More Than Six Minutes
Description: In participants with atrial fibrillation as evaluated by the LifestarAct III.
Time Frame: Week 2
Population: Due to software error, data could not be extracted for analysis for this outcome for all participants
Arm/Group | Cardiac Event Monitor
Number analyzed (Participants) | 0

5. Secondary Outcome: The Number of Participants With Frequent Premature Atrial Contractions
Description: More than 100 contraction during a 24 hour period as evaluated by the LifestarAct III.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Event Monitor
Number analyzed (Participants) | 85
Participants | 12

ADVERSE EVENTS:
Time Frame: Two weeks
Description: Only intervention related adverse events were collected for the study.
Arm/Group | Cardiac Event Monitor
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT02743520/Prot_SAP_000.pdf